CLINICAL TRIAL: NCT00898820
Title: Predictive Markers of Response to Pemetrexed (Companion Study to RC0524)
Brief Title: Tumor Response to Pemetrexed Disodium in Patients With Stage III or Stage IV Non-Small Cell Lung Cancer Enrolled in Clinical Trial MCCRC-RC0524
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Julian R. Molina, M.D., Ph.D., Mayo Clinic Cancer Center
Other Study IDs: RC0527; P30CA015083 (NIH); RC0527 (Other: Mayo Clinic Cancer Center & MCCRC); 06-002282 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving pemetrexed disodium may help doctors learn more about the effects of pemetrexed disodium on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This laboratory study is looking at blood samples from patients with stage III or stage IV non-small cell lung cancer enrolled in clinical trial MCCRC-RC0524 to determine the effect of pemetrexed disodium on cells.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the intracellular level of pemetrexed disodium (PD) polyglutamates as a measure of activity of PD transport and activation enzymes in patients with stage III or IV non-small cell lung cancer enrolled in clinical trial MCCRC-RC0524.

Secondary

* Assess polymorphisms and gene expression of PD target genes and genes encoding enzymes involved in the transport, activation, and inactivation of PD in these patients.
* Correlate haplotype-tagged single-nucleotide polymorphisms (htSNPs) and gene expression levels with intracellular levels of PD polyglutamates
* Correlate htSNPs and gene expression levels with toxicity and efficacy of PD.

OUTLINE: Blood is drawn prior to and 24 hours after day 1 of course 1 of pemetrexed disodium. DNA is extracted and genotyped for known polymorphisms in genes involved in the transport, activation, inactivation, and mechanism of action or resistance of pemetrexed disodium, including reduced folate carrier-1, multiresistance proteins (particularly MRP5), folate receptor, folypolyglutamate synthase, methylenetetrahydrofolate reductase (MTHFR), methionine synthase, methylthioadenosine phosphorylase, thymidylate synthase (TS), dihydrofolate reductase, and glycinamide ribonucleotide formyltransferase. Plasma and red blood cells are also processed for an intracellular polyglutamate assay for pemetrexed disodium by a high-performance liquid chromatography-based method.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled in clinical trial MCCRC-RC0524
* Willing to provide blood samples

PATIENT CHARACTERISTICS:

* No investigator site personnel directly affiliated with the study, or immediate family of investigator site personnel directly affiliated with the study

  * Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Not employed by Eli Lilly (i.e., employee, temporary contract worker, or designee responsible for conducting the study)

  * Immediate family of Eli Lilly employees allowed, but may not participate at an Eli Lilly facility

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Activity of pemetrexed disodium (PD) transport and activation enzymes as measured by intracellular content of PD polyglutamates

SECONDARY OUTCOMES:
Polymorphisms and gene expression of PD target genes (RFC-1, MRP, folate receptor, FPGS, methylenetetrahydrofolate reductase, methionine synthase, methylthioadenosine phosphorylase, TS, DHFR, GARFT)
Polymorphisms and gene expression of genes encoding enzymes involved in the transport, activation, and inactivation of PD
Correlation of haplotype-tagged single-nucleotide polymorphisms (htSNPs) and gene expression levels with intracellular levels of PD polyglutamates
Correlation of htSNPs and gene expression levels with toxicity and efficacy of PD

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, MD, PhD, Study Chair — Mayo Clinic; Elizabeth A. Johnson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States